CLINICAL TRIAL: NCT03067909
Title: THE Management of AntiThrOMbotic therApy in Patients Undergoing Electrophysiological Device Surgery: Italian NatiOnal Multicenter Observational REgistry (HEMATOMA NO MORE)
Brief Title: Antithrombotic Therapy in Patients Undergoing CIED Surgery - HEMATOMA NO MORE Registry
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Responsible Party: Principal Investigator, Valerio Zacà, Principal Investigator, Cardiology Consultant, Arrhythmology Unit, Cardiothoracic and Vascular Department, Azienda Ospedaliera Universitaria Senese
Other Study IDs: HNM_V1
Record Dates: First submitted 2017-02-25; First posted 2017-03-01 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Device Related Infection; Antithrombotic Drugs; Cardiac Arrhythmia; Surgery--Complications; Hematoma
MeSH Terms: conditions — Prosthesis-Related Infections; Arrhythmias, Cardiac; Hematoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing CIED surgery: Patients with standard indications to CIED implantations/replacements receiving concomitant antithrombotic therapy (either or both antiplatelet agents and/or anticoagulants).
  Interventions: Other: CIED surgery

INTERVENTIONS:
Other: CIED surgery

SUMMARY:
Hundreds of thousands patients undergo implantation or replacement of cardiac implantable electronic devices (CIEDs) annually in Europe, and up to 50% of these subjects receive antiplatelet agents or oral anticoagulants. Antithrombotic therapy increases the risk of developing pocket hematoma which in turn is associated with an increased risk of potentially fatal device-related infections when clinically significant. Aim of the registry is to retrospectively (pilot local registry in Tuscany) and prospectively (multicenter national registry in Italy) investigate the different strategies for the management of antithrombotic therapy and the related complication rates (1-month and 12-months) in patients undergoing CIED surgery in a real-world setting. The registry will also provide data on the economic impact of different management strategies and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with standard indications to CIED surgery being treated with antiplatelet agents and/or anticoagulants (any commercially available device or approved and marketed drug can be included).
* Patients able to provide written informed consent
* Patients willing to attend the planned follow-up visits

Exclusion Criteria:

* Patient with life expectancy less than 12 months as per investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients taking antithrombotic therapy undergoing CIED surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1450 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Clinically significant pocket hematoma | One month
  Post-procedural hematoma resulting in prolonged hospitalization and/or requiring interruption of antithrombotic therapy and/or requiring further surgery and/or requiring transfusion

SECONDARY OUTCOMES:
Non-clinically significant pocket hematoma | One month
  Post-procedural hematoma not meeting diagnostic criteria for clinically significant
Hemorrhagic complications other than pocket hematoma | One month
  Hemothorax, cardiac tamponade, pericardial effusion, intracranial hemorrhage
Thromboembolic complications | Twelve months
  Transient ischemic attack, ischemic stroke, deep venous thrombosis, pulmonary embolism, systemic embolic event, acute myocardial infarction, prosthetic cardiac valve thrombosis
All cause death | Twelve months
CIED-related infection | Twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Valerio Zacà, MD, Principal Investigator — AOU Senese
Locations (1):
- AOU Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available on demand to other researchers.

REFERENCES:
- [Background] Zaca V, Breschi M, Mandorli A, Panchetti L, Ricciardi G, Viani S, Notarstefano P. Rationale, study design, and pilot phase of tHE Management of AntiThrOMbotic therApy (HEMATOMA) in patients undergoing electrophysiological device surgery: Italian National Multicenter Observational REgistry. J Cardiovasc Med (Hagerstown). 2017 Nov;18(11):897-899. doi: 10.2459/JCM.0000000000000534. PMID 28594654
- [Background] V Zaca', A Angeletti, C Baiocchi, M Bertini, M Biffi, P Busacca, M Iori, M Mezzetti, M Nesti, P Notarstefano; P3213 Real-world periprocedural management of antithrombotic therapy in patients undergoing electrophysiological device surgery: preliminary results of the HEMATOMA NO MORE, European Heart Journal, Volume 39, Issue suppl_1, 1 August 2018, ehy563.P3213, https://doi.org/10.1093/eurheartj/ehy563.P3213